CLINICAL TRIAL: NCT01711463
Title: A Randomized, Double-blind, Placebo-controlled, Four-way Crossover Study to Evaluate and Compare the Pharmacodynamics and Pharmacokinetics of Fluticasone Furoate /Vilanterol in Different Dose Combination (50/25mcg, 100/25mcg and 200/25mcg) After Single and Repeat Dose Administration From a Novel Dry Powder Device in Healthy Chinese Subjects
Brief Title: Relovair PD PK in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 115199
Record Dates: First submitted 2012-08-30; First posted 2012-10-22 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: Pharmacodynamics; Fluticasone furoate (FF); novel dry powder device; Safety and tolerability; vilanterol(VI); Healthy Chinese subjects; Pharmacokinetics
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/VI (Experimental): 50/25 mcg, 100/25 mcg or 200/25 mcg
  Interventions: Drug: Fluticasone Furoate/Vilanterol
- Placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol — 50/25 or 100/25 or 200/25 mcg inhaled once daily for 7 days in each treatment period.
  Arms: FF/VI
Drug: Placebo — Placebo inhaled once daily for 7 days in each treatment period.
  Arms: Placebo

SUMMARY:
In this study, fluticasone furoate (FF) and vilanterol (VI) in different dose combinations (50/25mcg, 100/25mcg and 200/25mcg) will be administered from a single dry powder device to evaluate the PD, PK, safety and tolerability of the combination in healthy Chinese subjects. The information gathered will be used as a support of the clinical development program of the fixed dose combination of FF/VI inhalation powder in Chinese population.

DETAILED DESCRIPTION:
This is a single centre, double-blind, placebo-controlled, four-way cross over, randomized, single and repeat dose study. A total of 16 healthy subjects aged 18-45 years will be randomised with the aim of achieving at least 10 evaluable subjects to each treatment period. The primary objective is to evaluate the systemic steroid PD effects (serum cortisol 24 hour weighted mean on Day 7) of FF and systemic ß-adrenergic PD effects (ECG maximum QTcF 0-4h and whole blood potassium 0-4h in Day 1 and Day 7) of VI; the secondary objectives are aimed to evaluate the PK, safety and tolerability of FF/VI inhalation powder after a single and repeat dose administration.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy male or female between 18 and 45 years of age inclusive.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with blood pressure values outside the normal range [systolic (90-139 mmHg) and diastolic (50-89 mmHg)] and subjects with ECG findings suggestive of a previous MI should always be excluded from enrollment.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].

Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.

* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until completion of the follow-up visit.
* Body weight >= 50 kg and BMI within the range 19 - 24 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* No significant abnormality on 12-lead ECG at screening, including the following specific requirements:

Ventricular rate >= 45 beats per minute; PR interval <=210msec; No pathological Q waves; QRS interval to be >= 60msec and <=120msec; The waveforms must enable the QT interval to be clearly defined; QTc interval must be < 450msec (QTcF; machine or manual reading) based on a single ECG value, or an average from three ECGs obtained over a brief recording period.

* Subjects who are current non-smokers, who have not used any tobacco products in the 12 month period preceding the screening visit, and have a pack history of <=5 pack years.
* Subjects who are able to use the inhalation device satisfactorily.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen or on admission to the Unit.
* A positive urinary cotinine test at screening or on admission to the Unit.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a 285mL glass of full strength beer or 425mL schooner of light beer or 1 (30mL) measure of spirits or 1 glass (100mL) of wine (NHMRC Guidelines [NHMRC, 2001]).
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components (magnesium stearate and lactose etc.) or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of milk protein allergy.
* History of any adverse reaction including immediate or delayed hypersensitivity to any ICS, β2-agonist or sympathomimetic drug.
* Blood donation or sampled as a study subject within three months preceding the first dose of study drug and blood donation during the entire study.
* Pregnant females as determined by positive urine pregnancy test at screening or prior to dosing.
* Lactating females.
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* The subject has taken oral corticosteroids less than 8 weeks before the screening visit.
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2013-06-04 (Actual); Study Completion 2013-06-04 (Actual)

PRIMARY OUTCOMES:
Systemic steroid PD effects | Day 7
  Serum cortisol
Systemic ß-adrenergic PD effects | Day 1 and Day 7
  Maximum QTcF 0-4h and whole blood potassium

SECONDARY OUTCOMES:
Plasma concentrations and derived PK parameters for FF/VI | Pre-dose, 5 min, 15 min, 30 min, 1h, 1.5h, 2h, 4h post dose on Day 1 and pre-dose, 5 min, 15 min, 30 min, 1h, 1.5h, 2h, 4h, 6h, 8h, 12h and 24h post dose on Day 7 and 8.
  Single dose: Cmax, tmax, t1/2, AUC(0-t) (AUC from zero to the last quantifiable timepoint) and AUC(0-t') (AUC from zero to the last common quantifiable timepoint in the dose group). Repeat dose: FF: Cmax, tmax, t1/2, AUC(0-t) and AUC(0-t'), Ro and RCmax, Css_min and AUCss , Css_av, DF; VI: Cmax, tmax, t1/2, AUC(0-t) and AUC(0-t')
Vital signs | Screening Visit, Day 1, Day 7 and Follow-up Visit
  blood pressure and heart rate
12-lead ECG | Screening Visit, Day 1, Day 7 and Follow-up Visit
  12-lead ECG
Laboratory tests | Screening Visit, Day 8 of treatment period 4 or early withdrawal Visit and/or follow-up Visit
  Clinical chemistry, hematology and urinalysis
Adverse events | From the start of dosing with investigational product and until the follow-up visit.
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 115199 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115199?search=study&search_terms=115199#rs
- Available data/document: Study Protocol: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115199 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register